CLINICAL TRIAL: NCT00381537
Title: Prediction of Childhood Epilepsy Outcome in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Child Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 99NR58
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2006-12-25 (Estimated); Status verified 2006-12

CONDITIONS: Epilepsy
Keywords: childhood epilepsy; Active childhood epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Phenobarbital; Carbamazepine

INTERVENTIONS:
Drug: phenobarbitone
Drug: carbamazepine

SUMMARY:
Randomised controlled trial of the use of phenobarbitone and carbamazepine in childhood epilepsy in Bangladesh with particular reference to behavioural side effects.

ELIGIBILITY:
Inclusion Criteria:

* Active epilepsy
* Aged 2-15 years

Exclusion Criteria:

* Excluded absence
* Myoclonic and malignant epilepsy syndromes
* Major motor and cognitive impairments
* Those currently receiving antiepilepsy drugs.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92

CONTACTS AND LOCATIONS:
Overall Officials: Brian Neville, Professor, Principal Investigator — Institute of Child Health; Selina Banu, Dr, Principal Investigator — Children's Hospital Dhaka (Shishu) Bangladesh.
Locations (2):
- Children's Hospital Dhaka (Shishu) Bangladesh., Sher-e-Bangla Nagar, Dhaka 1207, Bangladesh
- Institute of Child Health, London, United Kingdom

REFERENCES:
- [Derived] Banu SH, Jahan M, Koli UK, Ferdousi S, Khan NZ, Neville B. Side effects of phenobarbital and carbamazepine in childhood epilepsy: randomised controlled trial. BMJ. 2007 Jun 9;334(7605):1207. doi: 10.1136/bmj.39022.436389.BE. Epub 2006 Dec 4. PMID 17145735